CLINICAL TRIAL: NCT01007461
Title: A Phase 2, Randomized. Double-Blind, Dose-Escalation, Dose-Expansion, Placebo-Controlled, Multi-Center Study of IK-1001 to Evaluate Safety, Pharmacokinetics , and Proof-of-Concept Efficacy in Subjects With Acute ST-Segment Elevation Myocardial Infarction (STEMI) Undergoing Primary Percutaneous Coronary Intervention
Brief Title: IK-1001 (Sodium Sulfide (Na2S) for Injection) in Subjects With Acute ST-Segment Elevation Myocardial Infarction
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decision. Non-safety related
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: IK-1001-AMI-201
Record Dates: First submitted 2009-10-26; First posted 2009-11-04 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: ST-Segment Elevation Myocardial Infraction
Keywords: Acute Myocardial Infarction (AMI); STEMI; Acute ST-Segment Elevation Myocardial Infraction (STEMI)
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — sodium sulfide; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IK-1001 (Experimental): IK-1001 Sodium Sulfide (Na2S) for Injection
  Interventions: Drug: Sodium Sulfide (Na2S) for Injection
- Placebo (Placebo Comparator): 0.9% Sodium Chloride (NaCl)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium Sulfide (Na2S) for Injection — IK-1001 is Na2S administered as an isotonic solution for intravenous (IV) injection or continuous infusion. IK-1001 will be administered as a 3-hour continuous IV infusion started > 5 minutes but < 20 minutes (approximately) prior to coronary artery reperfusion.
  Other Names: IK-1001
  Arms: IK-1001
Drug: Placebo — 0.9% Sodium Chloride (NaCl) will be administered in the same manner as the experimental drug.
  Arms: Placebo

SUMMARY:
Myocardial Infarctions (MI) are commonly known as heart attacks. An ST-Segment Elevation Myocardial Infarction (STEMI) is a more severe type of heart attack. Myocardial Infarctions happen when a coronary artery is partially or fully blocked suddenly by a blood clot, causing damage to at least some of the heart muscle being supplied by that artery. In a STEMI, a blood clot completely blocks the coronary artery. This can result in damage to the heart muscle that is supplied by the affected artery. The purpose of the IK-1001 STEMI Study is to evaluate the safety and effectiveness of an investigational study drug (IK-1001). IK-1001 is being studied to determine if it is safe and if it can reduce the amount of damage caused to the heart from a STEMI. Potential subjects may be eligible if they have been diagnosed with a STEMI and undergo a primary percutaneous coronary intervention (PCI, a procedure where a blocked coronary artery is unblocked during a cardiac catheterization), as well as meet other entry criteria. Up to 446 men and women, aged 18-80, will participate in this study at about 50 medical sites around the world. Study participation will last for about six months. Subjects will receive the study drug through an intravenous catheter over three hours during their PCI procedure. Subjects will be monitored in the hospital for approximately three to four days after the PCI. There are three follow-up visits at one, three and six months after the PCI with the study investigator after discharge from the hospital.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, dose-escalation, dose-expansion, double-blind, placebo-controlled, multi-center study that will evaluate safety, PK, and POC efficacy in subjects with acute STEMI undergoing PCI.

The study will be conducted in two parts. Part 1 is the dose escalation portion of the study. A minimum of 24 evaluable subjects will be enrolled into Part 1 to receive either IK-1001 (n = 18) or placebo (n = 6). Each subject will receive a continuous infusion of study drug at one of three dose escalating levels of 0.5, 1.0, or 1.5 mg/kg/hr infusion for 3 hours. At each dose level, 8 subjects will be enrolled (6 will receive IK-1001 and 2 will receive placebo). Placebo will consist of commercially available normal saline (NS) [0.9% sodium chloride (NaCl)].

Treatment with study drug (either IK-1001 or placebo) will be initiated only after informed consent is obtained and STEMI diagnosis is made based on clinical and ECG findings. ECG criteria for STEMI diagnosis include:

* Subjects presenting with ≥ 30 minutes of ischemic chest pain but within 12 hours of symptom onset
* Subjects having persistent ST-segment elevation of ≥ 2 mm in at least 2 contiguous leads in ECG

All subjects who receive study drug and have a successful PCI (defined as subjects in whom Grade 3 reperfusion was achieved) will be followed up for safety and efficacy for up to 6 months post-PCI and study drug infusion. Study samples will be collected from all subjects over the first 4 days following PCI for determination of PK parameters of sulfide in blood and thiosulfate in plasma. In Part 1, subjects who do not undergo a PCI for any reason will have study drug discontinued, will be excluded from the efficacy assessments but will be followed up for safety for 7 days, and will be replaced with a new subject.

Part 2 of the study will be an expansion of the highest safe continuous infusion dose evaluated in Part 1. Part 2 aims to further evaluate safety and establish POC efficacy at this dosing level. Initially, up to 190 eligible subjects will be randomized to receive either IK-1001 or placebo at a 1:1 ratio. Two interim analyses (IAs) will be done after 64 and 128 subjects complete the MI size evaluation at Day 4 (range 3 to 5 days), respectively. If there is a safety concern at any dose level, then enrollment in Part 2 will restart at the next lower safe dosing level determined from Part 1. If there is only an adequate or no efficacy signal at any dose level, then enrollment in Part 2 may restart at either an increased dose level (e.g., 1.75 mg/kg/hr for 3 hours) or at a longer duration of infusion (1.5 mg/kg/hr for 6 hours). A decision to stop the trial for safety, efficacy, or futility will be assessed at each IA. No more than 446 subjects will be enrolled in Part 2 of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Presentation to study hospital or institution with diagnosis of STEMI based on clinical and ECG findings (subject presented with ≥ 30 minutes of ischemic chest pain, within 12 hours of symptom onset, and has persistent ST-segment elevation of ≥ 2 mm ST-segment elevation in at least 2 contiguous leads in the ECG.
2. Age between 18 and 80 years (inclusive)
3. Signed Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved informed consent form

Exclusion Criteria:

1. Prior MI (as determined by subject history and/or ECG), cardiac surgery, or severe pericardial, congenital, cardiomyopathic, or valvular heart disease
2. Cardiac arrest within the past 28 days
3. Requirement for urgent cardiac surgery
4. Previous CABG surgery or PCI
5. Evidence of moderate or severe CHF (Killip Classes III and IV)
6. Any bradyarrhythmia that is expected to require a pacemaker through Day 4 (range 3 to 5 days), thus preventing the MRI
7. Unable to undergo a MRI (including disallowed metallic implants, unable to tolerate gadolinium contrast media, morbid obesity, or severe claustrophobia)
8. Subjects with past or current renal impairment requiring dialysis
9. Active or recent hemorrhage requiring an invasive procedure for evaluation or transfusion or hemorrhagic stroke within 6 weeks prior to presentation
10. Known or suspected aortic dissection
11. Subjects who have received treatment for asthma within the past 12 months
12. Prior history of pulmonary disease requiring chronic oxygen therapy
13. Females of childbearing potential
14. Body weight > 150 kg or Body Mass Index (BMI) > 40 kg/m2
15. Medical problem likely to preclude completion of the study
16. Use of investigational drugs or devices within 30 days prior to enrollment into the study
17. Any underlying medical or psychiatric condition that, in the opinion of the Investigator, makes the subject an unsuitable candidate for the study
18. Known food allergy to sulfite-containing foods and/or any drug allergies to drugs that contain sulfur

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Creatine Kinase, Muscle and Brain (CK-MB) Troponin T | Days 1 through 4, end of treatment

SECONDARY OUTCOMES:
12-Lead ECG | Study duration
Vital Signs | Study duration
Adverse Events | Study Duration
Cardiac magnetic resonance imaging (MRI) | Day 4, end of treatment